CLINICAL TRIAL: NCT00977067
Title: A Phase Ia, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of GDC-0152, an IAP Protein Antagonist, Administered Intravenously to Patients With Locally Advanced or Metastatic Malignancies
Brief Title: A Study of the Safety and Pharmacokinetics of GDC-0152, Administered Intravenously to Patients With Locally Advanced or Metastatic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early by the Sponsor for reasons unrelated to patient safety or anti-tumor activity.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAP4050g
Record Dates: First submitted 2009-09-12; First posted 2009-09-15 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Solid Cancers
Keywords: GDC0152; IAP; IAP Antagonist
MeSH Terms: interventions — GDC-0152

ARMS (1):
- A (Experimental)
  Interventions: Drug: GDC-0152

INTERVENTIONS:
Drug: GDC-0152 — Intravenous escalating dose

SUMMARY:
The study consists of two stages. In Stage 1, maximum tolerated dose (MTD) will be determined. In Stage 2, additional patients will be treated at the MTD of GDC-0152.

ELIGIBILITY:
Inclusion Criteria

* Histologically documented, incurable, locally advanced or metastatic solid malignancies, or non-Hodgkin's lymphoma (NHL) without leukemic phase
* Disease (either target or non-target lesions) that can be assessed by imaging studies and/or physical examination
* For patients with solid tumors or NHL without leukemic phase, disease progression on or after standard therapy, or a malignancy for which there is no standard therapy
* All prior therapy-related toxicities have recovered to baseline-grade toxicity with the exception of alopecia.
* Life expectancy of ≥ 60 days
* Resting oxygen saturation ≥ 92% on room air
* Agreement to use an effective form of contraception for the duration of the study

Exclusion Criteria

* History of central nervous system disease
* Chemotherapy, cancer hormonal therapy (except GnRH agonists), radiotherapy, or immunotherapy within 4 weeks prior to Day 1 (6 weeks for nitrosoureas or mitomycin)
* Use of any other investigational agent or device
* Major surgery or significant traumatic injury within 3 weeks prior to Day 1
* Pregnant or nursing
* Clinically significant cardiovascular disease, New York Heart Association (NYHA) Classification Grade 2 or greater congestive heart failure, a ventricular arrhythmia requiring medication within 1 year prior to Day 1, or NYHA Grade 2 or greater peripheral vascular disease on Day 1
* Known HIV infection
* Patients with ongoing inflammatory processes or a Grade ≥ 2 fever or Grade ≥ 2 fever-associated constitutional symptoms (including rigors/chills, sweating, and others determined by the investigator), or a clinically significant systemic infection within the last month
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications
* History of any chronic liver disease, active hepatic infection, or evidence of hepatic cirrhosis, or Grade ≥ 2 liver dysfunction.
* Baseline oxygen requirement or history of pulmonary fibrosis
* Any signs or symptoms Grade ≥ 2 by National Cancer Institute Common Terminology Criteria for Adverse Events, Version 3.0, at study entry except for alopecia, pain, asymptomatic Grade 2 diffusing capacity of the lung for carbon monoxide (at the discretion of the investigator) or where otherwise specified
* Patients who need to take a concomitant medication, dietary supplement, or food that is a known inhibitor/inducer of the CYP3A4/5 and/or the 2C8 metabolic pathway or that has a narrow therapeutic window and involves these enzymes for their metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities | Through study completion or early study discontinuation
Incidence, nature, and severity of adverse events | Through study completion or early study discontinuation

SECONDARY OUTCOMES:
Pharmacokinetic parameters of GDC-0152 (total plasma exposure, maximum plasma concentration, and total plasma clearance) | Through study completion or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Iris Chan, M.D., Ph.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Shin YG, Jones SA, Murakami SC, Budha N, Ware J, Wong H, Buonarati MH, Dean B, Hop CE. Validation and application of a liquid chromatography-tandem mass spectrometric method for the determination of GDC-0152 in human plasma using solid-phase extraction. Biomed Chromatogr. 2013 Jan;27(1):102-10. doi: 10.1002/bmc.2754. Epub 2012 May 24. PMID 22623056